CLINICAL TRIAL: NCT06356675
Title: A Single-arm Pilot Study of Tislelizumab Combined With Anlotinib in Patients With Advanced NSCLC With Driver-negative After Progression to Immunotherapy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Linzhu Zhai, professor of medicine，Deputy Director of Department of Radiotherapy, Oncology Center, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A single-arm pilot
Record Dates: First submitted 2024-03-25; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Advanced NSCLC
Keywords: Progress in first-line immunotherapy
MeSH Terms: interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Tislelizumab 200mg iv D1+anlotinib(12mg D1-12)
  Interventions: Drug: Tislelizumab; Drug: Anlotinib

INTERVENTIONS:
Drug: Tislelizumab — 200mg iv D1 Q3W
Drug: Anlotinib — Anlotinib 12mg D1-12 Q3W

SUMMARY:
Immune resistance after treatment, there is no standard treatment, one of the most important and the most effective measures is immune to combination therapy。Targeted angiogenesis therapy has always been the focus of research on the treatment of NSCLC patients with progressive disease after immunotherapy. From the mechanism of action, angiogenesis and immunosuppression are interrelated processes.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary participation in clinical research; Fully understand and Informed the study and sign the Informed Consent Form (ICF); Be willing to follow and be able to complete all trial procedures;
2. age of 18-75 years old (including boundary value), regardless of gender;
3. Pathologically confirmed locally advanced, metastatic non-small cell lung cancer (NSCLC), including squamous non-small cell lung cancer and non-squamous non-small cell lung cancer. Patients with non-squamous non-small cell lung cancer should exclude known EGFR mutation or ALK gene rearrangement.
4. patients with resistance to first-line PD-(L)1 inhibitors combined with chemotherapy;
5. patients with tumor response of CR/PR/SD after at least one first-line immunotherapy;
6. Subjects' ECOG PS score was 0-1 (including boundary value);
7. Patients had to have ≥1 measurable lesion (according to RECIST1.1 criteria).
8. predicted survival time ≥6 months;

Exclusion Criteria:

1. Frontline treatment with anlotinib, anti-angiogenic macromolecular monoclonal antibody or other small molecule TKI drugs;
2. central lung cancer with large blood vessel invasion;
3. patients with any signs or history of bleeding that may affect treatment according to the investigator's judgment; Patients with bleeding events ≥CTCAE grade 3, unhealed wounds, ulcers, or fractures within 4 weeks before the first dose of study drug;
4. hemoptysis > 50ml/d;
5. inability to swallow capsules or diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, gastric or small bowel resection, bariatric surgery, inflammatory bowel disease, partial or complete intestinal obstruction;
6. Poorly controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg)
7. other known malignant tumors that are developing or require active treatment;
8. Currently participating or has participated in the clinical research of other drugs;
9. interstitial lung disease or (non-infectious) pneumonia requiring steroid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The rate of tumor shrinkage reached 30% at least .including part reponse and complete response

SECONDARY OUTCOMES:
progression free survival time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  the time from initiation of treatment to disease progression or death as assessed by the treating physicians in the study (investigator-assessed).
over survival time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to18 months
  the time from initiation of treatment to death as assessed by the treating physicians in the study (investigator-assessed).
disease control rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  assessment of tumor the rate of the tumor harvest control including CR.PR and SD
safety including any grade adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  The adverse event type and the proportion of AE during the progress of disease treatment